CLINICAL TRIAL: NCT05546515
Title: Safety and Efficacy of Suvorexant for Opioid/Stimulant Co-use Among Individuals in Treatment for Opioid Use Disorder (OUD)
Brief Title: Suvorexant for Opioid/Stimulant Co-use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00341328
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; Stimulant Use Disorder
Keywords: Orexin receptor antagonist; Suvorexant; Cocaine; Opioid; Opiate; Heroin; Fentanyl; Nonmedical opioid use; Methadone; Buprenorphine; Suboxone; Polysubstance use; Co-use; Substance-related disorders; Narcotic-related disorders; Chemically-induced disorders; Sleep; Stress; Opioid-related disorders; Stimulant-related disorders; Cocaine use disorder
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Narcotic-Related Disorders; Chemically-Induced Disorders | interventions — suvorexant; Orexin Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research pharmacy will manage all randomization and blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suvorexant (Active Comparator): 20mg Suvorexant
  Interventions: Drug: Suvorexant (dual orexin receptor antagonist)
- Placebo (Placebo Comparator): Placebo oral capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant (dual orexin receptor antagonist) — Participants will be prescribed up to 30 days of SUVO.
  Arms: Suvorexant
Drug: Placebo — Participants will be prescribed up to 30 days of placebo medication.
  Arms: Placebo

SUMMARY:
This study will evaluate whether Suvorexant 20mg reduces drug use and craving, and improves sleep and stress among persons with co-occurring opioid use disorder and stimulant use disorder.

DETAILED DESCRIPTION:
This between-subjects, double-blinded, randomized controlled pilot study will recruit patients who are receiving methadone or buprenorphine treatment for OUD and are using cocaine. Participants will be randomly assigned to receive up to 30-days of Suvorexant (SUVO) or placebo. They will visit the clinic regularly to provide urine drug screens and complete questionnaires and will wear a device that can measure their sleep parameters. We expect that relative to persons who receive placebo, individuals who receive SUVO will 1) be less likely to screen positive for cocaine and/or opioids on urine drug screens, 2) will report lower drug craving, 3) will have longer total sleep time, 4) will report fewer insomnia symptoms, and 5) will report overall lower stress than persons who receive placebo. We also expect that patients will not have side effects from SUVO. These preliminary data will inform whether this FDA-approved medication may help patients stop co-using opioids and stimulants, which can be scaled up to reduce public health consequences related to co-use.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65,
2. Meet criteria for stimulant use disorder, based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR)
3. Currently receiving methadone or buprenorphine treatment for OUD and considered to be stable on current dose for at least 30 days
4. Willingness to engage with study protocol
5. Use of birth control (as appropriate)

Exclusion criteria:

1. Psychiatric or medical conditions that are judged by the investigators to interfere with participation or that are contraindicated for use with SUVO
2. Pregnant or breastfeeding
3. Current use of benzodiazepines, tranquilizers, or other schedule IV sleep medications
4. Moderate or severe substance use disorder other than opioid or stimulant use disorder
5. SUVO consumption in the last 30 days
6. Use of medications that are contraindicated with the study
7. Past 30-day suicidal behavior
8. Use of continuous positive airway pressure (CPAP) device for sleep apnea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ellis, Ph.D., Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Behavioral Pharmacology Research Unit at the Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 41 individuals attended a screening visit. Of the 20 individuals enrolled (i.e., initially determined as eligible to be scheduled for randomization), 5 declined enrollment and 2 no longer met criteria at the randomization visit and were not randomized.
  A total of 13 individuals were randomized. 12 of these individuals completed the study, one individual did not complete.
Period: Overall Study
Arm/Group | Suvorexant | Placebo
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.67 (9.54) | 49.14 (9.19) | 46.62 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: score on a scale] — Total score (sum of items). Total possible range = 0-28. Higher scores reflect greater insomnia symptoms.
  score on a scale | 15.67 (6.71) | 12.29 (9.62) | 13.84 (8.25)
Total Sleep Time (TST) [Mean (Standard Deviation); unit: minutes] — Self-reported total sleep time. Higher scores reflect a longer total sleep time. (Range = 180-540 minutes) Population: Two participants (one in each group) do not have data collected on this scale at baseline
  minutes
    number analyzed (Participants) | 5 | 6 | 11
    (all) | 394 (104.31) | 385 (120.62) | 389.09 (107.93)
Opioid Craving Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — Total possible score = 0-100, Higher scores reflect higher opioid craving.
  units on a scale | 39.43 (23.90) | 33.77 (34.22) | 36.38 (28.85)
Cocaine Craving VAS, [Mean (Standard Deviation); unit: units on a scale] — Total possible score = 0-100, Higher scores reflect higher cocaine craving.
  units on a scale | 44.27 (28.16) | 45.49 (30.28) | 44.92 (28.09)
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — Total score (sum of items). Total possible range = 0-40. Higher scores reflect greater perceived stress.
  units on a scale | 18.83 (10.34) | 19.14 (10.67) | 19 (10.07)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use: Proportion of Positive Urine Drug Screens (UDS)
Description: Opioid use (measured via uranalysis for qualitative opioid assay) other than prescribed methadone or buprenorphine at scheduled study visits up to 30 days post-randomization (yes vs. no)
Time Frame: Up to 30 days post-randomization
Population: One participant in the placebo group discontinued following randomization and did not have data collected.
Measure: Mean (Standard Deviation); unit: Proportion of urine drug screens
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 6 | 6
Proportion of urine drug screens | 0.83 (0.41) | 0.67 (0.52)

2. Primary Outcome: Cocaine Use: Proportion of Positive UDS Screens
Description: Cocaine use (measured via uranalysis for qualitative cocaine assay) at scheduled study visits up to 30 days post-randomization.
Time Frame: Up to 30 days post-randomization
Population: One participant in the placebo group discontinued following randomization and did not have data collected.
Measure: Mean (Standard Deviation); unit: Proportion of urine drug screens
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 6 | 6
Proportion of urine drug screens | 0.83 (0.41) | 0.97 (0.07)

3. Secondary Outcome: Insomnia Severity Regression Slope
Description: Regression slope of Insomnia Severity Index (ISI) scores over scheduled study visits through 30 days post-randomization. Total score range between 0-28 (absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28). Higher score worse insomnia.
Time Frame: Up to 30 days post-randomization
Population: One participant in the placebo group discontinued following randomization and did not have data collected, leaving six participants in each group.
Measure: Number (95% Confidence Interval); unit: score on a scale/day
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale/day | -0.55 [-1.02 to -0.08] | -0.16 [-0.64 to 0.33]

4. Secondary Outcome: Total Sleep Time (TST) Regression Slope
Description: Regression slope of TST scores over scheduled study visits up to 30 days post-randomization.
Time Frame: Up to 30 days post-randomization
Population: Two participants did not have baseline data on TST and could not be included in the analysis. One additional participant in the placebo group discontinued following randomization and did not have data collected.
Measure: Number (95% Confidence Interval); unit: score on a scale/day
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale/day | 11.68 [-4.35 to 27.7] | 9.37 [-7.93 to 26.7]

5. Secondary Outcome: Opioid Craving Visual Analog Scale (VAS) Regression Slope
Description: Regression slope of opioid craving VAS scores over scheduled study visits through 30 days post-randomization. Score range 0-10 with higher score indicating worse craving.
Time Frame: Up to 30 days post-randomization
Population: One participant in the placebo group discontinued following randomization and did not have data collected.
Measure: Number (95% Confidence Interval); unit: score on a scale/day
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale/day | -1.76 [-5.65 to 2.12] | -1.46 [-5.43 to 2.51]

6. Secondary Outcome: Cocaine Craving Visual Analog Scale (VAS) Regression Slope
Description: Regression slope of cocaine craving VAS scores over scheduled study visits through 30 days post-randomization. Score range 0-10 with higher score indicating worse craving.
Time Frame: Up to 30 days post-randomization
Population: One participant in the placebo group discontinued following randomization and did not have data collected.
Measure: Number (95% Confidence Interval); unit: score on a scale/day
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale/day | -0.60 [-2.66 to 1.46] | -0.71 [-2.86 to 1.44]

7. Secondary Outcome: Perceived Stress Scale Regression Slope
Description: Regression slope of Perceived Stress Scale (PSS) scores over scheduled study visits through 30 days post-randomization. Total score range 0 to 40, with higher scores indicating worse perceived stress.
Time Frame: Up to 30 days post-randomization
Population: One participant in the placebo group discontinued following randomization and did not have data collected.
Measure: Number (95% Confidence Interval); unit: score on a scale/day
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale/day | -0.19 [-0.62 to 0.24] | 0.19 [-0.26 to 0.64]

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up, up to 30 days
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 6/6 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suvorexant (N=6) | Placebo (N=7)
Edema (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Hypertension (Cardiac disorders) | 4 | 5
Tachycardia (Cardiac disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Appetite increased (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Toothache (General disorders) | 2 | 0
Drowsiness (Nervous system disorders) | 4 | 0
Skin rash (Skin and subcutaneous tissue disorders) | 2 | 0 — Irritation from actigraph

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT05546515/Prot_SAP_000.pdf